CLINICAL TRIAL: NCT02861534
Title: A Randomized Parallel-Group, Placebo-Controlled, Double-Blind, Event-Driven, Multi-Center Pivotal Phase III Clinical Outcome Trial of Efficacy and Safety of the Oral sGC Stimulator Vericiguat in Subjects With Heart Failure With Reduced Ejection Fraction (HFrEF) - VerICiguaT GlObal Study in Subjects With Heart Failure With Reduced EjectIon FrAction (VICTORIA)
Brief Title: A Study of Vericiguat in Participants With Heart Failure With Reduced Ejection Fraction (HFrEF) (MK-1242-001)
Acronym: VICTORIA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Bayer (Industry); Canadian VIGOUR Centre (Other); Duke Clinical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1242-001; 2016-000671-25 (EudraCT Number); MK-1242-001 (Other: Merck Protocol Number)
Record Dates: First submitted 2016-08-05; First posted 2016-08-10 (Estimated); Results first posted 2020-06-29 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Heart Failure; Chronic Heart Failure With Reduced Ejection Fraction
MeSH Terms: conditions — Heart Failure | interventions — vericiguat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vericiguat (Experimental): Participants receive a starting dose of 2.5 mg of vericiguat taken orally once daily with food, on a background of HF standard of care. The vericiguat dose will be uptitrated to 5 mg and to 10 mg.
  Interventions: Drug: Vericiguat
- Placebo (Placebo Comparator): Participants receive a starting matching placebo dose of 2.5 mg taken orally once daily with food, on a background of HF standard of care. The matching placebo dose will be uptitrated to 5 mg and to 10 mg.
  Interventions: Drug: Placebo for vericiguat

INTERVENTIONS:
Drug: Vericiguat — 2.5, 5.0, or 10.0 mg orally once daily
  Other Names: MK-1242
  Arms: Vericiguat
Drug: Placebo for vericiguat — 2.5, 5.0, or 10.0 mg orally once daily
  Arms: Placebo

SUMMARY:
This is a randomized, placebo-controlled, parallel-group, multi-center, double-blind, event driven study of vericiguat (MK-1242) in participants with heart failure with reduced ejection fraction (HFrEF). The primary hypothesis is vericiguat (MK-1242) is superior to placebo in increasing the time to first occurrence of the composite of cardiovascular (CV) death or heart failure (HF) hospitalization in participants with HFrEF.

ELIGIBILITY:
Inclusion Criteria:

* History of chronic HF (New York Heart Association [NYHA] Class II-IV) on standard therapy before qualifying HF decompensation
* Previous HF hospitalization within 6 months prior to randomization or intravenous (IV) diuretic treatment for HF (without hospitalization) within 3 months.
* Brain natriuretic peptide (BNP) levels: sinus rhythm-≥ 300 pg/mL; atrial fibrillation-≥ 500 pg/mL and N-terminal pro-Brain Natriuretic Peptide (NT-proBNP) levels: sinus rhythm- ≥ 1000 pg/mL; atrial fibrillation - ≥ 1600 pg/mL within 30 days prior to randomization
* Left ventricular ejection fraction (LVEF) of <45% assessed within 12 months prior to randomization by any method
* If female, is not of reproductive potential or agrees to avoid becoming pregnant while receiving study drug and for 14 days after the last dose of study drug by complying with one of the following: practice abstinence from heterosexual activity or use (or have her partner use) acceptable contraception during heterosexual activity.

Exclusion Criteria:

* Clinically unstable at the time of randomization as defined by either the administration of any IV treatment within 24 hours prior to randomization, and/or systolic blood pressure (SBP) <100 mmHg or symptomatic hypotension
* Current or anticipated use of long-acting nitrates or nitric oxide (NO) donors including isosorbide dinitrate, isosorbide 5-mononitrate, pentaerythritol tetranitrate, nicorandil or transdermal nitroglycerin (NTG) patch, and molsidomine
* Current or anticipated use of phosphodiesterase type 5 (PDE5) inhibitors such as vardenafil, tadalafil, and sildenafil
* Current use or anticipated use of a soluble guanylate cyclase (sGC) stimulator such as riociguat
* Known allergy or sensitivity to any sGC stimulator
* Awaiting heart transplantation (United Network for Organ Sharing Class 1A / 1B or equivalent), receiving continuous IV infusion of an inotrope, or has/anticipates receiving an implanted ventricular assist device
* Primary valvular heart disease requiring surgery or intervention, or is within 3 months after valvular surgery or intervention
* Hypertrophic obstructive cardiomyopathy
* Acute myocarditis, amyloidosis, sarcoidosis, Takotsubo cardiomyopathy
* Post-heart transplant cardiomyopathy
* Tachycardia-induced cardiomyopathy and/or uncontrolled tachyarrhythmia
* Acute coronary syndrome (unstable angina, non-ST elevation myocardial infarction [NSTEMI], or ST elevation myocardial infarction [(STEMI]) or coronary revascularization (coronary artery bypass grafting [CABG] or percutaneous coronary intervention [PCI]) within 60 days, or indication for coronary revascularization at time of randomization
* Symptomatic carotid stenosis, transient ischemic attack (TIA) or stroke within 60 days
* Complex congenital heart disease
* Active endocarditis or constrictive pericarditis
* Estimated glomerular filtration rate (eGFR) <15 mL/min/1.73 m2 or chronic dialysis
* Severe hepatic insufficiency such as with hepatic encephalopathy
* Malignancy or other non-cardiac condition limiting life expectancy to <3 years
* Require continuous home oxygen for severe pulmonary disease
* Current alcohol and/or drug abuse
* Participated in another interventional clinical study and treatment with another investigational product ≤30 days prior to randomization or plans to participate in any other trial/investigation during the duration of this study
* Mental or legal incapacitation and is unable to provide informed consent
* Immediate family member (e.g., spouse, parent/legal guardian, sibling or child) who is involved with this study
* Interstitial Lung Disease
* Is pregnant or breastfeeding or plans to become pregnant or to breastfeed during the course of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5050 (Actual)
Dates: Start 2016-09-20 (Actual); Primary Completion 2019-06-18 (Actual); Study Completion 2019-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mahesh J. Patel, MD, Study Director — Merck Sharp & Dohme LLC; Paul W. Armstrong, MD, Study Chair — Canadian VIGOUR Centre - University of Alberta; Christopher M. O'Connor, MD, Principal Investigator — Inova Heart and Vascular Institute; Burkert Pieske, MD, Principal Investigator — Charité University Medicine and German Heart Center

IPD SHARING:
Plan to Share IPD: Yes
https://thecvc.ca/victoria/data-sharing/

REFERENCES:
- [Result] Pieske B, Patel MJ, Westerhout CM, Anstrom KJ, Butler J, Ezekowitz J, Hernandez AF, Koglin J, Lam CSP, Ponikowski P, Roessig L, Voors AA, O'Connor CM, Armstrong PW; VICTORIA Study Group. Baseline features of the VICTORIA (Vericiguat Global Study in Subjects with Heart Failure with Reduced Ejection Fraction) trial. Eur J Heart Fail. 2019 Dec;21(12):1596-1604. doi: 10.1002/ejhf.1664. Epub 2019 Dec 9. PMID 31820546
- [Derived] Shah P, Zheng Y, Pieske B, Melenovsky V, Lam CSP, Sliwa K, Butler J, Ezekowitz JA, deFilippi CR, O'Connor CM, Sandhu RK, Roessig L, Tromp J, Westerhout CM, Voors AA, Armstrong PW; VICTORIA Study Group. Phenomapping in Heart Failure With Reduced Ejection Fraction to Identify Subpopulations With High Residual Risk: A VICTORIA Substudy. Circ Heart Fail. 2025 Oct 8:e013166. doi: 10.1161/CIRCHEARTFAILURE.125.013166. Online ahead of print. PMID 41058565
- [Derived] Khan MS, Butler J, Young R, Lewis BS, Escobedo J, Refsgaard J, Reyes E, Roessig L, Blaustein RO, Lam CSP, Voors AA, Ponikowski P, Anstrom KJ, Armstrong PW; VICTORIA Study Group. Vericiguat and Cardiovascular Outcomes in Heart Failure by Baseline Diabetes Status: Insights From the VICTORIA Trial. JACC Heart Fail. 2024 Oct;12(10):1750-1759. doi: 10.1016/j.jchf.2024.05.007. Epub 2024 Jun 26. PMID 38934967
- [Derived] Mentz RJ, Stebbins A, Butler J, Chiang CE, Ezekowitz JA, Hernandez AF, Hilkert R, Lam CSP, McDonald K, O'Connor CM, Pieske B, Ponikowski P, Roessig L, Sweitzer NK, Voors AA, Anstrom KJ, Armstrong PW; VICTORIA Study Group. Recurrent Hospitalizations and Response to Vericiguat in Heart Failure and Reduced Ejection Fraction. JACC Heart Fail. 2024 May;12(5):839-846. doi: 10.1016/j.jchf.2023.12.005. Epub 2024 Feb 14. PMID 38363272
- [Derived] Chew DS, Li Y, Bigelow R, Cowper PA, Anstrom KJ, Daniels MR, Davidson-Ray L, Hernandez AF, O'Connor CM, Armstrong PW, Mark DB; VICTORIA Study Group. Cost-Effectiveness of Vericiguat in Patients With Heart Failure With Reduced Ejection Fraction: The VICTORIA Randomized Clinical Trial. Circulation. 2023 Oct 3;148(14):1087-1098. doi: 10.1161/CIRCULATIONAHA.122.063602. Epub 2023 Sep 6. PMID 37671551
- [Derived] Lam CSP, Pina IL, Zheng Y, Bonderman D, Pouleur AC, Saldarriaga C, Pieske B, Blaustein RO, Nkulikiyinka R, Westerhout CM, Armstrong PW; VICTORIA Study Group. Age, Sex, and Outcomes in Heart Failure With Reduced EF: Insights From the VICTORIA Trial. JACC Heart Fail. 2023 Sep;11(9):1246-1257. doi: 10.1016/j.jchf.2023.06.020. Epub 2023 Aug 9. PMID 37565973
- [Derived] Armstrong PW, Zheng Y, Lund LH, Butler J, Troughton RW, Emdin M, Lam CSP, Ponikowski P, Blaustein RO, O'Connor CM, Roessig L, Voors AA, Ezekowitz JA, Westerhout CM; VICTORIA Study Group. Evolution of NT-proBNP During Prerandomization Screening in VICTORIA: Implications for Clinical Outcomes and Efficacy of Vericiguat. Circ Heart Fail. 2023 Oct;16(10):e010661. doi: 10.1161/CIRCHEARTFAILURE.123.010661. Epub 2023 Jul 28. PMID 37503602
- [Derived] Ezekowitz JA, McMullan CJ, Westerhout CM, Pina IL, Lopez-Sendon J, Anstrom KJ, Hernandez AF, Lam CSP, O'Connor CM, Pieske B, Ponikowski P, Roessig L, Voors AA, Koglin J, Armstrong PW, Butler J; VICTORIA Study Group. Background Medical Therapy and Clinical Outcomes From the VICTORIA Trial. Circ Heart Fail. 2023 Sep;16(9):e010599. doi: 10.1161/CIRCHEARTFAILURE.123.010599. Epub 2023 Jul 7. PMID 37417824
- [Derived] Felker GM, North R, Mulder H, Jones WS, Anstrom KJ, Patel MJ, Butler J, Ezekowitz JA, Lam CSP, O'Connor CM, Roessig L, Hernandez AF, Armstrong PW; VICTORIA Study Group. Classification of Heart Failure Events by Severity: Insights From the VICTORIA Trial. J Card Fail. 2023 Aug;29(8):1113-1120. doi: 10.1016/j.cardfail.2023.04.015. Epub 2023 Jun 17. PMID 37331690
- [Derived] Butler J, Zheng Y, Khan MS, Bonderman D, Lund LH, deFilippi CR, Blaustein RO, Ezekowitz JA, Freitas C, Hernandez AF, O'Connor CM, Voors AA, Westerhout CM, Lam CSP, Armstrong PW; VICTORIA Study Group. Ejection Fraction, Biomarkers, and Outcomes and Impact of Vericiguat on Outcomes Across EF in VICTORIA. JACC Heart Fail. 2023 May;11(5):583-592. doi: 10.1016/j.jchf.2022.12.014. Epub 2023 Apr 12. PMID 37137660
- [Derived] Armstrong PW, Zheng Y, Troughton RW, Lund LH, Zhang J, Lam CSP, Westerhout CM, Blaustein RO, Butler J, Hernandez AF, Roessig L, O'Connor CM, Voors AA, Ezekowitz JA; VICTORIA Study Group. Sequential Evaluation of NT-proBNP in Heart Failure: Insights Into Clinical Outcomes and Efficacy of Vericiguat. JACC Heart Fail. 2022 Sep;10(9):677-688. doi: 10.1016/j.jchf.2022.04.015. Epub 2022 Jul 6. PMID 36049817
- [Derived] Senni M, Lopez-Sendon J, Cohen-Solal A, Ponikowski P, Nkulikiyinka R, Freitas C, Vlajnic VM, Roessig L, Pieske B. Vericiguat and NT-proBNP in patients with heart failure with reduced ejection fraction: analyses from the VICTORIA trial. ESC Heart Fail. 2022 Dec;9(6):3791-3803. doi: 10.1002/ehf2.14050. Epub 2022 Jul 26. PMID 35880474
- [Derived] Senni M, Alemayehu WG, Sim D, Edelmann F, Butler J, Ezekowitz J, Hernandez AF, Lam CSP, O'Connor CM, Pieske B, Ponikowski P, Roessig L, Voors AA, Westerhout CM, McMullan C, Armstrong PW; VICTORIA Study Group. Efficacy and safety of vericiguat in patients with heart failure with reduced ejection fraction treated with sacubitril/valsartan: insights from the VICTORIA trial. Eur J Heart Fail. 2022 Sep;24(9):1614-1622. doi: 10.1002/ejhf.2608. Epub 2022 Jul 20. PMID 35791083
- [Derived] Butler J, Stebbins A, Melenovsky V, Sweitzer NK, Cowie MR, Stehlik J, Khan MS, Blaustein RO, Ezekowitz JA, Hernandez AF, Lam CSP, Nkulikiyinka R, O'Connor CM, Pieske BM, Ponikowski P, Spertus JA, Voors AA, Anstrom KJ, Armstrong PW; VICTORIA Study Group. Vericiguat and Health-Related Quality of Life in Patients With Heart Failure With Reduced Ejection Fraction: Insights From the VICTORIA Trial. Circ Heart Fail. 2022 Jun;15(6):e009337. doi: 10.1161/CIRCHEARTFAILURE.121.009337. Epub 2022 Jun 3. PMID 35656822
- [Derived] Lam CSP, Mulder H, Lopatin Y, Vazquez-Tanus JB, Siu D, Ezekowitz J, Pieske B, O'Connor CM, Roessig L, Patel MJ, Anstrom KJ, Hernandez AF, Armstrong PW; VICTORIA Study Group. Blood Pressure and Safety Events With Vericiguat in the VICTORIA Trial. J Am Heart Assoc. 2021 Nov 16;10(22):e021094. doi: 10.1161/JAHA.121.021094. Epub 2021 Nov 6. PMID 34743540
- [Derived] Ezekowitz JA, Zheng Y, Cohen-Solal A, Melenovsky V, Escobedo J, Butler J, Hernandez AF, Lam CSP, O'Connor CM, Pieske B, Ponikowski P, Voors AA, deFilippi C, Westerhout CM, McMullan C, Roessig L, Armstrong PW. Hemoglobin and Clinical Outcomes in the Vericiguat Global Study in Patients With Heart Failure and Reduced Ejection Fraction (VICTORIA). Circulation. 2021 Nov 2;144(18):1489-1499. doi: 10.1161/CIRCULATIONAHA.121.056797. Epub 2021 Aug 25. PMID 34432985
- [Derived] Ezekowitz J, Mentz RJ, Westerhout CM, Sweitzer NK, Givertz MM, Pina IL, O'Connor CM, Greene SJ, McMullan C, Roessig L, Hernandez AF, Armstrong PW. Participation in a Heart Failure Clinical Trial: Perspectives and Opportunities From the VICTORIA Trial and VICTORIA Simultaneous Registry. Circ Heart Fail. 2021 Sep;14(9):e008242. doi: 10.1161/CIRCHEARTFAILURE.120.008242. Epub 2021 Aug 19. PMID 34407626
- [Derived] Mentz RJ, Mulder H, Mosterd A, Sweitzer NK, Senni M, Butler J, Ezekowitz JA, Lam CSP, Pieske B, Ponikowski P, Voors AA, Anstrom KJ, Armstrong PW, O'connor CM, Hernandez AF; VICTORIA Study Group. Clinical Outcome Predictions for the VerICiguaT Global Study in Subjects With Heart Failure With Reduced Ejection Fraction (VICTORIA) Trial. J Card Fail. 2021 Jun 24:S1071-9164(21)00206-2. doi: 10.1016/j.cardfail.2021.05.016. Online ahead of print. PMID 34217593
- [Derived] Mentz RJ, Mulder H, Mosterd A, Sweitzer NK, Senni M, Butler J, Ezekowitz JA, Lam CSP, Pieske B, Ponikowski P, Voors AA, Anstrom KJ, Armstrong PW, O'Connor CM; VICTORIA Study Group. Clinical Outcome Predictions for the VerICiguaT Global Study in Subjects With Heart Failure With Reduced Ejection Fraction (VICTORIA) Trial: VICTORIA Outcomes Model. J Card Fail. 2021 May 26:S1071-9164(21)00206-2. doi: 10.1016/j.cardfail.2021.05.016. Online ahead of print. PMID 34216757
- [Derived] Lam CSP, Giczewska A, Sliwa K, Edelmann F, Refsgaard J, Bocchi E, Ezekowitz JA, Hernandez AF, O'Connor CM, Roessig L, Patel MJ, Pieske B, Anstrom KJ, Armstrong PW; VICTORIA Study Group. Clinical Outcomes and Response to Vericiguat According to Index Heart Failure Event: Insights From the VICTORIA Trial. JAMA Cardiol. 2021 Jun 1;6(6):706-712. doi: 10.1001/jamacardio.2020.6455. PMID 33185650
- [Derived] Ezekowitz JA, O'Connor CM, Troughton RW, Alemayehu WG, Westerhout CM, Voors AA, Butler J, Lam CSP, Ponikowski P, Emdin M, Patel MJ, Pieske B, Roessig L, Hernandez AF, Armstrong PW. N-Terminal Pro-B-Type Natriuretic Peptide and Clinical Outcomes: Vericiguat Heart Failure With Reduced Ejection Fraction Study. JACC Heart Fail. 2020 Nov;8(11):931-939. doi: 10.1016/j.jchf.2020.08.008. Epub 2020 Oct 7. PMID 33039447
- [Derived] Armstrong PW, Pieske B, Anstrom KJ, Ezekowitz J, Hernandez AF, Butler J, Lam CSP, Ponikowski P, Voors AA, Jia G, McNulty SE, Patel MJ, Roessig L, Koglin J, O'Connor CM; VICTORIA Study Group. Vericiguat in Patients with Heart Failure and Reduced Ejection Fraction. N Engl J Med. 2020 May 14;382(20):1883-1893. doi: 10.1056/NEJMoa1915928. Epub 2020 Mar 28. PMID 32222134
- [Derived] Armstrong PW, Roessig L, Patel MJ, Anstrom KJ, Butler J, Voors AA, Lam CSP, Ponikowski P, Temple T, Pieske B, Ezekowitz J, Hernandez AF, Koglin J, O'Connor CM. A Multicenter, Randomized, Double-Blind, Placebo-Controlled Trial of the Efficacy and Safety of the Oral Soluble Guanylate Cyclase Stimulator: The VICTORIA Trial. JACC Heart Fail. 2018 Feb;6(2):96-104. doi: 10.1016/j.jchf.2017.08.013. Epub 2017 Oct 11. PMID 29032136

RESULTS

PARTICIPANT FLOW:
Groups:
- Vericiguat: Participants received a starting dose of 2.5 mg of vericiguat taken orally once daily with food, on a background of heart failure (HF) standard of care. The vericiguat dose was uptitrated to 5 mg and to 10 mg.
- Placebo: Participants received a starting matching placebo dose of 2.5 mg taken orally once daily with food, on a background of HF standard of care. The matching placebo dose was uptitrated to 5 mg and to 10 mg.
Period: Overall Study
Arm/Group | Vericiguat | Placebo
Started | 2526 | 2524
Treated | 2519 | 2515
Completed | 1952 | 1937
Not Completed | 574 | 587
Not completed — Death | 541 | 552
Not completed — Lost to Follow-up | 14 | 14
Not completed — Site Terminated by Sponsor | 4 | 3
Not completed — Withdrawal by Subject | 15 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vericiguat | Placebo | Total
Number analyzed (Participants) | 2526 | 2524 | 5050
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.5 (12.2) | 67.2 (12.2) | 67.3 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 605 | 603 | 1208
  Male | 1921 | 1921 | 3842
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 24 | 28 | 52
  Asian | 571 | 561 | 1132
  Native Hawaiian or Other Pacific Islander | 3 | 11 | 14
  Black or African American | 123 | 126 | 249
  White | 1621 | 1618 | 3239
  More than one race | 183 | 180 | 363
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Secondary Outcome: Time to the First Occurrence of CV Death
Description: Time to First Occurrence of CV Death was analyzed using a one-sided stratified log-rank test. Randomized participants without a CV death at the time of analysis were censored at their last available information, the date of their non-CV death, or the primary analysis database cutoff date of 18-June-2019, whichever occurred first. A CEC reviewed and adjudicated the endpoint events. A time-to-event methodology was used to evaluate the results; the incidence rate of participants with an event (number of participants with an event per 100 participant-years at risk) is provided.
Time Frame: Up to approximately 33 months (through primary analysis database cutoff date of 18-June-2019)
Population: All randomized participants
Measure: Number; unit: Parts w/ event per 100 part-yrs at risk
Groups:
- Vericiguat: Participants received a starting dose of 2.5 mg of vericiguat taken orally once daily with food, on a background of HF standard of care. The vericiguat dose was uptitrated to 5 mg and to 10 mg.
Arm/Group | Vericiguat | Placebo
Number analyzed (Participants) | 2526 | 2524
Parts w/ event per 100 part-yrs at risk | 12.9 | 13.9
Statistical Analysis 1: Comparison: Vericiguat vs Placebo; Test type: Superiority; p = 0.269, Cox proportional hazard model; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.81 to 1.06]

2. Secondary Outcome: Time to the First Occurrence of HF Hospitalization
Description: Time to the First Occurrence of HF Hospitalization was analyzed using a one-sided stratified log-rank test. Randomized participants without any HF hospitalization at the time of analysis were censored at their last available information, the date of their death, or the primary analysis database cutoff date of 18-June-2019, whichever occurred first. A CEC reviewed and adjudicated the endpoint events. A time-to-event methodology was used to evaluate the results; the incidence rate of participants with an event (number of participants with an event per 100 participant-years at risk) is provided.
Time Frame: Up to approximately 33 months (through primary analysis database cutoff date of 18-June-2019)
Population: All randomized participants
Measure: Number; unit: Parts w/ event per 100 part-yrs at risk
Arm/Group | Vericiguat | Placebo
Number analyzed (Participants) | 2526 | 2524
Parts w/ event per 100 part-yrs at risk | 25.9 | 29.1
Statistical Analysis 1: Comparison: Vericiguat vs Placebo; Test type: Superiority; p = 0.048, Cox proportional hazard model; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.81 to 1.00]

3. Primary Outcome: Time to First Occurrence of Composite Endpoint of Cardiovascular (CV) Death or Heart Failure (HF) Hospitalization
Description: Time to First Occurrence of Composite Endpoint of CV Death or HF Hospitalization was analyzed using a one-sided stratified log-rank test. Randomized participants without any HF hospitalization or CV death event at the time of analysis were censored at their last available information, the date of their non-CV death, or the primary analysis database cutoff date of 18-June-2019, whichever occurred first. A clinical events committee (CEC) reviewed and adjudicated the endpoint events. A time-to-event methodology was used to evaluate the results; the incidence rate of participants with an event (number of participants with an event per 100 participant-years at risk) is provided.
Time Frame: Up to approximately 33 months (through primary analysis database cutoff date of 18-June-2019)
Population: All randomized participants
Measure: Number; unit: Parts w/ event per 100 part-yrs at risk
Arm/Group | Vericiguat | Placebo
Number analyzed (Participants) | 2526 | 2524
Parts w/ event per 100 part-yrs at risk | 33.6 [41.5 to 46.4] | 37.8 [44.4 to 49.4]
Statistical Analysis 1: Comparison: Vericiguat vs Placebo; Test type: Superiority; p = 0.019, Cox proportional hazard model; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.82 to 0.98]

4. Secondary Outcome: Time to Total HF Hospitalizations (Including First and Recurrent Events)
Description: Time to Total HF Hospitalizations (including first and recurring) was analyzed using an Andersen-Gill model. Randomized participants without any HF hospitalization at the time of analysis were censored at their last available information, the date of their death, or the primary analysis database cutoff date of 18-June-2019, whichever occurred first. A CEC reviewed and adjudicated the endpoint events. A time-to-event methodology was used to evaluate the results; the incidence rate of participants with an event (number of participants with an event per 100 participant-years of follow-up) is provided.
Time Frame: Up to approximately 33 months (through primary analysis database cutoff date of 18-June-2019)
Population: All randomized participants
Measure: Number; unit: Parts w/ event per 100 part-yrs
Arm/Group | Vericiguat | Placebo
Number analyzed (Participants) | 2526 | 2524
Parts w/ event per 100 part-yrs | 38.3 | 42.4
Statistical Analysis 1: Comparison: Vericiguat vs Placebo; Test type: Superiority; p = 0.023, Andersen-Gill model; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.84 to 0.99]

5. Secondary Outcome: Time to First Occurrence of Composite Endpoint of All-Cause Mortality or HF Hospitalization
Description: Time to First Occurrence of Composite Endpoint of All-Cause Mortality or HF Hospitalization was analyzed using a one-sided stratified log-rank test. Randomized participants without any all-cause mortality event or HF hospitalization at the time of analysis were censored at their last available information or the primary analysis database cutoff date of 18-June-2019, whichever occurred first. A CEC reviewed and adjudicated the endpoint events. A time-to-event methodology was used to evaluate the results; the incidence rate of participants with an event (number of participants with an event per 100 participant-years at risk) is provided.
Time Frame: Up to approximately 33 months (through primary analysis database cutoff date of 18-June-2019)
Population: All randomized participants
Measure: Number; unit: Parts w/ event per 100 part-yrs at risk
Arm/Group | Vericiguat | Placebo
Number analyzed (Participants) | 2526 | 2524
Parts w/ event per 100 part-yrs at risk | 35.9 | 40.1
Statistical Analysis 1: Comparison: Vericiguat vs Placebo; Test type: Superiority; p = 0.021, Cox proportional hazard model; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.83 to 0.98]

6. Secondary Outcome: Time to All-Cause Mortality
Description: Time to All-Cause Mortality was analyzed using a one-sided stratified log-rank test. Randomized participants without any all-cause mortality event at the time of analysis were censored at their last available information or the primary analysis database cutoff date of 18-June-2019, whichever occurred first. A CEC reviewed and adjudicated the endpoint events. A time-to-event methodology was used to evaluate the results: the incidence rate of participants with an event (number of participants with an event per 100 participant-years at risk) is provided.
Time Frame: Up to approximately 33 months (through primary analysis database cutoff date of 18-June-2019)
Population: All randomized participants
Measure: Number; unit: Parts w/ event per 100 part-yrs at risk
Arm/Group | Vericiguat | Placebo
Number analyzed (Participants) | 2526 | 2524
Parts w/ event per 100 part-yrs at risk | 16.0 | 16.9
Statistical Analysis 1: Comparison: Vericiguat vs Placebo; Test type: Superiority; p = 0.377, Cox proportional hazard model; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.84 to 1.07]

7. Secondary Outcome: Number of Participants Who Experienced One or More Adverse Events
Description: An adverse event (AE) is any untoward medical occurrence in a study participant administered a pharmaceutical product that does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not related to the medicinal product.
Time Frame: Up to approximately 33 months (through primary analysis database cutoff date of 18-June-2019)
Population: All randomized participants who received at least 1 dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Vericiguat | Placebo
Number analyzed (Participants) | 2519 | 2515
Participants | 2027 | 2036

8. Secondary Outcome: Number of Participants Who Discontinued Treatment Due to an Adverse Event
Description: as for outcome 7
Time Frame: Up to approximately 33 months (through primary analysis database cutoff date of 18-June-2019)
Population: All randomized participants who received at least 1 dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Vericiguat | Placebo
Number analyzed (Participants) | 2519 | 2515
Participants | 167 | 158

9. Secondary Outcome: Percentage of Participants Who Experienced Symptomatic Hypotension
Description: Study participants were monitored for symptomatic hypotension, an event of clinical interest, and results were reported.
Time Frame: Up to approximately 33 months (through primary analysis database cutoff date of 18-June-2019)
Population: All randomized participants who received at least 1 dose of study treatment
Measure: Number; unit: Percentage of participants
Arm/Group | Vericiguat | Placebo
Number analyzed (Participants) | 2519 | 2515
Percentage of participants | 9.1 | 7.9
Statistical Analysis 1: Comparison: Vericiguat vs Placebo; Test type: Other; p = 0.121, Miettinen & Nurminen method; Difference in Percentage = 1.2, 95% CI 2-sided [-0.3 to 2.8]

10. Secondary Outcome: Percentage of Participants Who Experienced Syncope
Description: Study participants were monitored for syncope, an event of clinical interest, and results were reported.
Time Frame: Up to approximately 33 months (through primary analysis database cutoff date of 18-June-2019)
Population: All randomized participants who received at least 1 dose of study treatment
Measure: Number; unit: Percentage of participants
Arm/Group | Vericiguat | Placebo
Number analyzed (Participants) | 2519 | 2515
Percentage of participants | 4.0 | 3.5
Statistical Analysis 1: Comparison: Vericiguat vs Placebo; Test type: Other; p = 0.303, Miettinen & Nurminen method; Difference in Percentage = 0.6, 95% CI 2-sided [-0.5 to 1.6]

ADVERSE EVENTS:
Time Frame: Up to approximately 35 months (through Last Subject Last Visit date of 02-Sept-2019)
Description: Serious Adverse Events and Other Adverse Events: All randomized participants who received at least 1 dose of study treatment
  All-Cause Mortality: All randomized participants
Arm/Group | Vericiguat | Placebo
All-Cause Mortality (participants affected / at risk) | 553/2526 | 561/2524
Serious Adverse Events (participants affected / at risk) | 852/2519 | 897/2515
Other Adverse Events (participants affected / at risk) | 958/2519 | 925/2515
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vericiguat (N=2519) | Placebo (N=2515)
Anaemia (Blood and lymphatic system disorders) | 41 (50) | 24 (25)
Anaemia of chronic disease (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Bicytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Blood loss anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Bone marrow failure (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hypocoagulable state (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 3 (3) | 2 (2)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Normocytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
Splenic infarction (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 4 (4)
Acute myocardial infarction (Cardiac disorders) | 5 (6) | 5 (5)
Angina pectoris (Cardiac disorders) | 9 (10) | 8 (9)
Angina unstable (Cardiac disorders) | 2 (2) | 7 (13)
Aortic valve calcification (Cardiac disorders) | 1 (1) | 0 (0)
Aortic valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 3 (3) | 3 (3)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 14 (15) | 29 (31)
Atrial flutter (Cardiac disorders) | 6 (7) | 7 (7)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Atrial thrombosis (Cardiac disorders) | 0 (0) | 2 (2)
Atrioventricular block (Cardiac disorders) | 2 (2) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 2 (2)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 1 (1)
Bradyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 3 (3) | 3 (3)
Bundle branch block left (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac arrest (Cardiac disorders) | 3 (3) | 3 (3)
Cardiac asthma (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 82 (88) | 116 (128)
Cardiac failure acute (Cardiac disorders) | 2 (2) | 4 (4)
Cardiac failure chronic (Cardiac disorders) | 5 (5) | 10 (10)
Cardiac failure congestive (Cardiac disorders) | 13 (13) | 25 (25)
Cardiac perforation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac ventricular thrombosis (Cardiac disorders) | 2 (2) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 4 (4) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 8 (8) | 4 (4)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 1 (1)
Cardiorenal syndrome (Cardiac disorders) | 3 (3) | 2 (2)
Cardiovascular disorder (Cardiac disorders) | 1 (1) | 0 (0)
Cardiovascular insufficiency (Cardiac disorders) | 1 (1) | 0 (0)
Congestive cardiomyopathy (Cardiac disorders) | 3 (3) | 3 (3)
Coronary artery disease (Cardiac disorders) | 7 (8) | 3 (3)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 3 (4) | 2 (2)
Extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Heart valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Intracardiac thrombus (Cardiac disorders) | 0 (0) | 2 (2)
Ischaemic cardiomyopathy (Cardiac disorders) | 1 (1) | 2 (2)
Left ventricular dysfunction (Cardiac disorders) | 1 (1) | 1 (1)
Left ventricular failure (Cardiac disorders) | 0 (0) | 2 (2)
Mitral valve incompetence (Cardiac disorders) | 7 (7) | 5 (5)
Myocardial infarction (Cardiac disorders) | 6 (6) | 3 (3)
Myocardial ischaemia (Cardiac disorders) | 3 (3) | 2 (2)
Palpitations (Cardiac disorders) | 2 (2) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 2 (2) | 2 (2)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tachyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 2 (2) | 1 (1)
Ventricular dysfunction (Cardiac disorders) | 0 (0) | 2 (2)
Ventricular extrasystoles (Cardiac disorders) | 2 (2) | 2 (2)
Ventricular fibrillation (Cardiac disorders) | 9 (10) | 7 (9)
Ventricular tachycardia (Cardiac disorders) | 14 (18) | 27 (29)
Corneal dystrophy (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Gastrointestinal arteriovenous malformation (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Hydrocele (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Phimosis (Congenital, familial and genetic disorders) | 1 (1) | 1 (1)
Pyloric stenosis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 3 (3) | 7 (7)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 3 (4)
Basedow's disease (Endocrine disorders) | 1 (1) | 0 (0)
Carcinoid syndrome (Endocrine disorders) | 1 (1) | 0 (0)
Glucocorticoid deficiency (Endocrine disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 4 (4) | 1 (1)
Hypoparathyroidism secondary (Endocrine disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Blindness (Eye disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 9 (10) | 6 (8)
Diabetic retinopathy (Eye disorders) | 2 (2) | 1 (1)
Diplopia (Eye disorders) | 1 (1) | 0 (0)
Eye haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Eyelid ptosis (Eye disorders) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 1 (1) | 0 (0)
Macular cyst (Eye disorders) | 0 (0) | 1 (1)
Retinal artery thrombosis (Eye disorders) | 1 (1) | 0 (0)
Retinal haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Vitreous haemorrhage (Eye disorders) | 2 (2) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 4 (4)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 4 (5) | 3 (3)
Abdominal rigidity (Gastrointestinal disorders) | 1 (1) | 0 (0)
Alcoholic pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anorectal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 8 (10) | 4 (5)
Barrett's oesophagus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 2 (2) | 2 (2)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3) | 2 (2)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dental cyst (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 10 (10) | 7 (7)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulum intestinal (Gastrointestinal disorders) | 1 (1) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 3 (3)
Erosive oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastric perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastritis (Gastrointestinal disorders) | 4 (4) | 7 (7)
Gastritis erosive (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 12 (14) | 7 (7)
Gastrointestinal toxicity (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 4 (4)
Gingival bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 3 (3) | 2 (2)
Ileus (Gastrointestinal disorders) | 2 (2) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 2 (2) | 0 (0)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 (0) | 3 (3)
Incarcerated umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 11 (11) | 9 (9)
Inguinal hernia strangulated (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia, obstructive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal infarction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intra-abdominal haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ischaemic enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestinal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestinal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestinal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestinal ulcer perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 1 (2) | 4 (4)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Obstructive pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal achalasia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 2 (2) | 1 (1)
Pancreatitis chronic (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pancreatolithiasis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pneumatosis intestinalis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 4 (4) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0)
Subileus (Gastrointestinal disorders) | 0 (0) | 2 (2)
Umbilical hernia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (3) | 6 (6)
Vomiting (Gastrointestinal disorders) | 4 (4) | 2 (2)
Asthenia (General disorders) | 6 (6) | 6 (7)
Cardiac complication associated with device (General disorders) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 2 (2)
Chest pain (General disorders) | 10 (10) | 8 (14)
Device related thrombosis (General disorders) | 0 (0) | 1 (1)
Discomfort (General disorders) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 6 (6) | 1 (1)
Generalised oedema (General disorders) | 1 (1) | 0 (0)
Hernia (General disorders) | 1 (1) | 0 (0)
Impaired healing (General disorders) | 0 (0) | 1 (1)
Implant site erythema (General disorders) | 0 (0) | 1 (1)
Implant site haematoma (General disorders) | 2 (2) | 0 (0)
Implant site haemorrhage (General disorders) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 1 (1)
Medical device pain (General disorders) | 1 (1) | 0 (0)
Medical device site haematoma (General disorders) | 2 (2) | 0 (0)
Medical device site swelling (General disorders) | 0 (0) | 1 (1)
Medical device site thrombosis (General disorders) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 2 (2) | 4 (4)
Non-cardiac chest pain (General disorders) | 4 (4) | 7 (7)
Oedema (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 3 (3)
Physical deconditioning (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 3 (3) | 2 (2)
Sensation of foreign body (General disorders) | 1 (1) | 0 (0)
Strangulated hernia (General disorders) | 0 (0) | 1 (1)
Sudden cardiac death (General disorders) | 0 (0) | 1 (1)
UGT1A1 gene polymorphism (General disorders) | 0 (0) | 1 (1)
Vascular stent occlusion (General disorders) | 1 (1) | 0 (0)
Vascular stent stenosis (General disorders) | 1 (1) | 0 (0)
Vascular stent thrombosis (General disorders) | 0 (0) | 1 (1)
Acute hepatic failure (Hepatobiliary disorders) | 1 (1) | 3 (3)
Bile duct stone (Hepatobiliary disorders) | 2 (2) | 1 (1)
Biloma (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholangitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 4 (4) | 4 (4)
Cholecystitis acute (Hepatobiliary disorders) | 4 (4) | 6 (6)
Cholecystitis chronic (Hepatobiliary disorders) | 2 (2) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 4 (4) | 2 (2)
Cholestasis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Chronic hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 2 (2) | 1 (1)
Hepatic congestion (Hepatobiliary disorders) | 4 (4) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatitis acute (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatitis toxic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatocellular injury (Hepatobiliary disorders) | 2 (2) | 0 (0)
Ischaemic hepatitis (Hepatobiliary disorders) | 4 (4) | 2 (2)
Jaundice cholestatic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 2 (2) | 0 (0)
Liver injury (Hepatobiliary disorders) | 5 (5) | 2 (2)
Portosplenomesenteric venous thrombosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Amyloidosis (Immune system disorders) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 3 (3) | 2 (2)
Acinetobacter bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Amoebic dysentery (Infections and infestations) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 2 (2) | 1 (1)
Arteriovenous fistula site infection (Infections and infestations) | 0 (0) | 1 (1)
Atypical pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Bacterial sepsis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 10 (10) | 7 (7)
Bronchitis viral (Infections and infestations) | 2 (2) | 1 (1)
Campylobacter gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 25 (27) | 19 (20)
Cellulitis gangrenous (Infections and infestations) | 1 (1) | 0 (0)
Chest wall abscess (Infections and infestations) | 1 (1) | 0 (0)
Cholecystitis infective (Infections and infestations) | 0 (0) | 2 (2)
Chronic sinusitis (Infections and infestations) | 1 (1) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 2 (2) | 0 (0)
Complicated appendicitis (Infections and infestations) | 2 (2) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Cystitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 4 (4) | 2 (2)
Diabetic foot infection (Infections and infestations) | 1 (1) | 2 (2)
Diarrhoea infectious (Infections and infestations) | 1 (1) | 1 (1)
Disseminated tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 2 (2)
Endocarditis (Infections and infestations) | 4 (7) | 1 (1)
Enteritis infectious (Infections and infestations) | 1 (1) | 0 (0)
Enterobacter bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Enterococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Enterococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Enterocolitis viral (Infections and infestations) | 0 (0) | 1 (1)
Epididymitis (Infections and infestations) | 2 (2) | 0 (0)
Erysipelas (Infections and infestations) | 2 (2) | 6 (6)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Extradural abscess (Infections and infestations) | 1 (1) | 0 (0)
Eye infection bacterial (Infections and infestations) | 0 (0) | 1 (1)
Febrile infection (Infections and infestations) | 0 (0) | 1 (1)
Fungaemia (Infections and infestations) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 4 (4) | 4 (4)
Gas gangrene (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 16 (16) | 10 (10)
Gastroenteritis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis norovirus (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis salmonella (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Groin abscess (Infections and infestations) | 0 (0) | 2 (2)
H1N1 influenza (Infections and infestations) | 1 (1) | 0 (0)
Haematoma infection (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Implant site cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Implant site infection (Infections and infestations) | 3 (3) | 3 (3)
Infected bite (Infections and infestations) | 0 (0) | 1 (1)
Infected skin ulcer (Infections and infestations) | 2 (2) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 3 (3)
Infectious pleural effusion (Infections and infestations) | 1 (1) | 1 (1)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 (1) | 3 (3)
Influenza (Infections and infestations) | 11 (11) | 8 (8)
Intervertebral discitis (Infections and infestations) | 1 (1) | 1 (1)
Intestinal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Klebsiella sepsis (Infections and infestations) | 0 (0) | 1 (1)
Liver abscess (Infections and infestations) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 7 (8) | 4 (4)
Lower respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 10 (12) | 3 (3)
Measles (Infections and infestations) | 1 (1) | 0 (0)
Medical device site abscess (Infections and infestations) | 0 (0) | 1 (1)
Myocarditis infectious (Infections and infestations) | 1 (1) | 0 (0)
Necrotising fasciitis (Infections and infestations) | 2 (2) | 0 (0)
Nosocomial infection (Infections and infestations) | 1 (1) | 0 (0)
Ophthalmic herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 6 (6) | 6 (7)
Osteomyelitis acute (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis chronic (Infections and infestations) | 1 (1) | 0 (0)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0)
Parainfluenzae virus infection (Infections and infestations) | 1 (1) | 1 (1)
Parotid abscess (Infections and infestations) | 0 (0) | 1 (1)
Periodontitis (Infections and infestations) | 1 (1) | 1 (1)
Perirectal abscess (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1)
Peritonitis bacterial (Infections and infestations) | 2 (2) | 0 (0)
Pertussis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 104 (113) | 116 (127)
Pneumonia bacterial (Infections and infestations) | 3 (3) | 4 (4)
Pneumonia chlamydial (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia mycoplasmal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia streptococcal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia viral (Infections and infestations) | 1 (1) | 1 (1)
Postoperative wound infection (Infections and infestations) | 2 (2) | 1 (1)
Pseudomembranous colitis (Infections and infestations) | 0 (0) | 2 (2)
Psoas abscess (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 2 (2) | 3 (3)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis chronic (Infections and infestations) | 0 (0) | 1 (1)
Renal abscess (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 5 (5) | 4 (4)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1)
Salmonella bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 16 (16) | 25 (25)
Septic shock (Infections and infestations) | 11 (11) | 14 (14)
Serratia bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Skin bacterial infection (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 2 (4) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 2 (2) | 2 (2)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal skin infection (Infections and infestations) | 1 (1) | 0 (0)
Streptococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0)
Systemic candida (Infections and infestations) | 1 (1) | 0 (0)
Thrombophlebitis septic (Infections and infestations) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1)
Tracheobronchitis (Infections and infestations) | 2 (2) | 0 (0)
Tuberculous pleurisy (Infections and infestations) | 1 (1) | 0 (0)
Typhoid fever (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 11 (11) | 10 (10)
Ureter abscess (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 20 (23) | 16 (18)
Urosepsis (Infections and infestations) | 7 (8) | 0 (0)
Vestibular neuronitis (Infections and infestations) | 1 (1) | 2 (2)
Viral diarrhoea (Infections and infestations) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 2 (2) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 3 (3) | 0 (0)
West Nile viral infection (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 4 (4)
Wound sepsis (Infections and infestations) | 0 (0) | 2 (2)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Arterial bypass occlusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Asbestosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Bone fissure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Burns second degree (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Burns third degree (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Cardiac valve replacement complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Chest injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Coronary vascular graft stenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Costal cartilage fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 6 (6) | 5 (5)
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 (3) | 8 (8)
Femur fracture (Injury, poisoning and procedural complications) | 3 (3) | 12 (12)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
Heat illness (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 6 (6) | 3 (3)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb crushing injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 5 (5)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Penis injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haematuria (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural hypothyroidism (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Postoperative hypotension (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pubis fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sedation complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Snake bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Subdural haematoma (Injury, poisoning and procedural complications) | 6 (6) | 1 (1)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Suture related complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 6 (6)
Traumatic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic liver injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic ulcer (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Urinary retention postoperative (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular graft occlusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Vasoplegia syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Angiocardiogram (Investigations) | 1 (1) | 1 (1)
Anticoagulation drug level above therapeutic (Investigations) | 2 (2) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 2 (2)
Blood creatinine increased (Investigations) | 1 (1) | 1 (1)
Blood potassium increased (Investigations) | 1 (1) | 0 (0)
Blood sodium decreased (Investigations) | 1 (1) | 0 (0)
Blood urea increased (Investigations) | 0 (0) | 1 (1)
Bone density abnormal (Investigations) | 1 (1) | 0 (0)
Cardiac index abnormal (Investigations) | 1 (1) | 0 (0)
Cardiac stress test abnormal (Investigations) | 0 (0) | 1 (1)
Catheterisation cardiac (Investigations) | 1 (1) | 1 (1)
Cortisol decreased (Investigations) | 0 (0) | 1 (1)
Ejection fraction decreased (Investigations) | 0 (0) | 3 (3)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1) | 1 (1)
Heart rate irregular (Investigations) | 0 (0) | 1 (1)
Hepatic enzyme abnormal (Investigations) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 2 (2) | 2 (2)
Influenza A virus test positive (Investigations) | 0 (0) | 1 (1)
International normalised ratio increased (Investigations) | 1 (1) | 2 (2)
Liver function test abnormal (Investigations) | 1 (1) | 0 (0)
Liver function test increased (Investigations) | 1 (1) | 1 (1)
Occult blood positive (Investigations) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 1 (1)
Troponin increased (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 1 (1)
Weight increased (Investigations) | 0 (0) | 1 (1)
Cachexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 7 (7) | 12 (13)
Diabetes mellitus (Metabolism and nutrition disorders) | 5 (6) | 10 (11)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Diabetes with hyperosmolarity (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 4 (4) | 2 (2)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Gout (Metabolism and nutrition disorders) | 10 (12) | 12 (14)
Hyperammonaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 6 (6) | 4 (4)
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 13 (13) | 14 (14)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperosmolar state (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypochloraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 12 (13) | 9 (9)
Hypokalaemia (Metabolism and nutrition disorders) | 7 (8) | 7 (7)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 5 (5) | 5 (5)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Marasmus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 2 (2) | 4 (4)
Metabolic alkalosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Mineral metabolism disorder (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 5 (5) | 8 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 3 (3)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chondritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Enthesopathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 7 (9) | 6 (7)
Gouty tophus (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (2) | 5 (5)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spondylitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adrenal gland cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Angiocentric lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Benign gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 4 (4)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cutaneous T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatobiliary cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Inflammatory pseudotumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 4 (4)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to abdominal cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oropharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oropharyngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Polycythaemia vera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 5 (5)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Retroperitoneal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of head and neck (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Sweat gland tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour ulceration (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Waldenstrom's macroglobulinaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Altered state of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Autonomic neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Axonal neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Brain hypoxia (Nervous system disorders) | 1 (1) | 0 (0)
Brain injury (Nervous system disorders) | 2 (2) | 1 (1)
Brain oedema (Nervous system disorders) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 3 (3)
Cauda equina syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral artery embolism (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral artery stenosis (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 2 (2)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 3 (3) | 6 (6)
Cerebrovascular disorder (Nervous system disorders) | 1 (1) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 1 (1)
Coma (Nervous system disorders) | 1 (1) | 0 (0)
Dementia (Nervous system disorders) | 2 (2) | 0 (0)
Dementia Alzheimer's type (Nervous system disorders) | 0 (0) | 2 (2)
Diabetic neuropathy (Nervous system disorders) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 6 (6) | 2 (2)
Dizziness postural (Nervous system disorders) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 0 (0) | 2 (2)
Encephalopathy (Nervous system disorders) | 0 (0) | 2 (2)
Facial paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 2 (2) | 2 (2)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Lumbar radiculopathy (Nervous system disorders) | 2 (2) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 2 (2)
Myelopathy (Nervous system disorders) | 1 (1) | 0 (0)
Myoclonus (Nervous system disorders) | 0 (0) | 2 (2)
Neuropathy peripheral (Nervous system disorders) | 2 (2) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Post stroke epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 4 (4) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 2 (2) | 2 (2)
Spinal cord compression (Nervous system disorders) | 0 (0) | 1 (1)
Status epilepticus (Nervous system disorders) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 43 (45) | 33 (35)
Tension headache (Nervous system disorders) | 1 (1) | 0 (0)
Toxic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 2 (2) | 2 (2)
Vascular dementia (Nervous system disorders) | 0 (0) | 1 (1)
Vertebrobasilar insufficiency (Nervous system disorders) | 1 (1) | 0 (0)
Device battery issue (Product Issues) | 1 (1) | 4 (4)
Device dislocation (Product Issues) | 0 (0) | 2 (3)
Device failure (Product Issues) | 0 (0) | 1 (1)
Device ineffective (Product Issues) | 0 (0) | 1 (1)
Device malfunction (Product Issues) | 1 (1) | 4 (4)
Lead dislodgement (Product Issues) | 1 (2) | 0 (0)
Alcohol abuse (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 2 (2)
Delirium (Psychiatric disorders) | 0 (0) | 3 (4)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Drug use disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 2 (2)
Panic attack (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 66 (69) | 51 (53)
Azotaemia (Renal and urinary disorders) | 0 (0) | 1 (1)
Bladder cyst (Renal and urinary disorders) | 1 (1) | 0 (0)
Bladder mass (Renal and urinary disorders) | 0 (0) | 1 (1)
Calculus bladder (Renal and urinary disorders) | 2 (2) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 40 (42) | 31 (31)
Costovertebral angle tenderness (Renal and urinary disorders) | 0 (0) | 1 (1)
End stage renal disease (Renal and urinary disorders) | 2 (2) | 1 (1)
Haematuria (Renal and urinary disorders) | 3 (3) | 7 (7)
Nephritis (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephropathy (Renal and urinary disorders) | 3 (3) | 1 (1)
Nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal artery stenosis (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal cyst (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 24 (25) | 30 (31)
Renal impairment (Renal and urinary disorders) | 6 (6) | 7 (7)
Renal infarct (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal mass (Renal and urinary disorders) | 1 (1) | 0 (0)
Urate nephropathy (Renal and urinary disorders) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 2 (2) | 0 (0)
Urethral stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 2 (2) | 2 (2)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 8 (8)
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 7 (7)
Asthma (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 4 (6)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchial haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 38 (51) | 30 (50)
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 7 (7)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 13 (15)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 6 (6)
Pulmonary haematoma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (4)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5)
Rhinitis hypertrophic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Tonsillar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Henoch-Schonlein purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Neurodermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 5 (5) | 9 (14)
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Aortic aneurysm repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Arrhythmia prophylaxis (Surgical and medical procedures) | 0 (0) | 1 (1)
Cardiac pacemaker replacement (Surgical and medical procedures) | 0 (0) | 1 (1)
Cardiac rehabilitation therapy (Surgical and medical procedures) | 1 (1) | 0 (0)
Cardiac resynchronisation therapy (Surgical and medical procedures) | 2 (2) | 7 (7)
Cardiovascular event prophylaxis (Surgical and medical procedures) | 1 (1) | 4 (4)
Cardioversion (Surgical and medical procedures) | 1 (3) | 0 (0)
Central venous catheter removal (Surgical and medical procedures) | 0 (0) | 1 (1)
Gastrectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Implantable defibrillator insertion (Surgical and medical procedures) | 5 (5) | 2 (2)
Implantable defibrillator removal (Surgical and medical procedures) | 1 (1) | 0 (0)
Implantable defibrillator replacement (Surgical and medical procedures) | 1 (1) | 0 (0)
Inguinal hernia repair (Surgical and medical procedures) | 1 (1) | 0 (0)
Intraocular lens implant (Surgical and medical procedures) | 0 (0) | 1 (1)
Leg amputation (Surgical and medical procedures) | 1 (1) | 0 (0)
Nephroprotective therapy (Surgical and medical procedures) | 0 (0) | 1 (1)
Therapeutic procedure (Surgical and medical procedures) | 1 (1) | 0 (0)
Toe operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 1 (1) | 2 (2)
Aortic dissection (Vascular disorders) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 1 (1) | 1 (1)
Arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1)
Bleeding varicose vein (Vascular disorders) | 1 (1) | 2 (2)
Circulatory collapse (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Diabetic vascular disorder (Vascular disorders) | 1 (1) | 0 (0)
Dry gangrene (Vascular disorders) | 0 (0) | 1 (1)
Extremity necrosis (Vascular disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 4 (4) | 2 (3)
Haemorrhagic vasculitis (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 5 (5) | 4 (4)
Hypertensive crisis (Vascular disorders) | 1 (1) | 5 (5)
Hypotension (Vascular disorders) | 33 (34) | 44 (45)
Hypovolaemic shock (Vascular disorders) | 2 (2) | 0 (0)
Iliac artery occlusion (Vascular disorders) | 1 (1) | 0 (0)
Intermittent claudication (Vascular disorders) | 2 (2) | 1 (1)
Ischaemia (Vascular disorders) | 1 (1) | 0 (0)
Lymphorrhoea (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 6 (6) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 6 (6) | 11 (12)
Peripheral artery occlusion (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery stenosis (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Peripheral embolism (Vascular disorders) | 1 (1) | 2 (2)
Peripheral ischaemia (Vascular disorders) | 2 (2) | 3 (3)
Peripheral vascular disorder (Vascular disorders) | 4 (6) | 3 (3)
Peripheral venous disease (Vascular disorders) | 1 (1) | 0 (0)
Shock (Vascular disorders) | 1 (1) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 2 (2)
Thrombophlebitis (Vascular disorders) | 1 (1) | 2 (2)
Varicose vein (Vascular disorders) | 1 (1) | 0 (0)
Varicose vein ruptured (Vascular disorders) | 1 (1) | 0 (0)
Vascular occlusion (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vericiguat (N=2519) | Placebo (N=2515)
Anaemia (Blood and lymphatic system disorders) | 165 (181) | 134 (139)
Cardiac failure (Cardiac disorders) | 160 (219) | 157 (221)
Diarrhoea (Gastrointestinal disorders) | 127 (141) | 120 (136)
Nasopharyngitis (Infections and infestations) | 126 (153) | 131 (163)
Hyperkalaemia (Metabolism and nutrition disorders) | 112 (124) | 138 (167)
Dizziness (Nervous system disorders) | 169 (195) | 152 (169)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 127 (161) | 132 (158)
Hypotension (Vascular disorders) | 369 (487) | 331 (437)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-20): https://cdn.clinicaltrials.gov/large-docs/34/NCT02861534/Prot_SAP_000.pdf